CLINICAL TRIAL: NCT02275481
Title: A Comparative Effectiveness and Safety Study of Arformoterol Tartrate Inhalation Solution and Tiotropium Bromide on Re-hospitalization in Chronic Obstructive Pulmonary Disease (COPD) Subjects
Brief Title: A Study of Arformoterol Tartrate Inhalation Solution and Tiotropium Bromide on Re-hospitalization in Chronic Obstructive Pulmonary Disease (COPD) Subjects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEP091-402
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive pulmonary disease; COPD; Emphysema; Chronic bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic | interventions — Formoterol Fumarate; Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BROVANA (Experimental): Arformoterol tartrate inhalation solution 15 mcg (BROVANA) will be administered BID (morning and evening, approximately 12 hours between doses) using a standard jet nebulizer with a face mask or mouthpiece connected to an air compressor
  Interventions: Drug: Arformoterol tartrate inhalation solution
- SPIRIVA (Active Comparator): Tiotropium 18 mcg (SPIRIVA) will be administered QD (morning) via the HandiHaler®.
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Arformoterol tartrate inhalation solution — Arformoterol tartrate inhalation solution 15 mcg (BROVANA) will be administered BID (morning and evening, approximately 12 hours between doses) using a standard jet nebulizer with a face mask or mouthpiece connected to an air compressor
  Other Names: BROVANA
  Arms: BROVANA
Drug: Tiotropium — Tiotropium 18 mcg (SPIRIVA) will be administered QD (morning) via the HandiHaler®.
  Other Names: SPIRIVA
  Arms: SPIRIVA

SUMMARY:
This is a randomized, open-label, parallel group, multicenter, outpatient study in COPD subjects who are discharged from the hospital due to a COPD exacerbation. Subjects who meet the eligibility criteria will be randomized to 1 of 2 treatments: arformoterol tartrate inhalation solution (BROVANA) 15 mcg twice daily (BID) or tiotropium bromide (SPIRIVA) 18 mcg once daily (QD), each given for 90 days.

DETAILED DESCRIPTION:
This is a randomized, open-label, parallel group, multicenter, outpatient study in COPD subjects who are discharged from the hospital following a COPD exacerbation. Subjects who meet the eligibility criteria will be randomized to 1 of 2 treatments. Arformoterol tartrate inhalation solution 15 mcg (BROVANA) will be administered BID (morning and evening, approximately 12 hours between doses) using a standard jet nebulizer with a face mask or mouthpiece connected to an air compressor. Tiotropium 18 mcg (SPIRIVA) will be administered QD (morning) via the HandiHaler®.

Study medications will be dispensed to the subject at Visit 1. The objective of the study is to determine the comparative effectiveness of arformoterol and tiotropium on re-hospitalization and to assess safety in Chronic Obstructive Pulmonary Disease (COPD) subjects recovering from hospitalization for an acute exacerbation.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥ 55 years-old are eligible for study participation if they have a physician-assessed diagnosis of COPD, have been discharged from the hospital due to a COPD exacerbation, and at least 1 of the following:

   1. Subject has had 1 or more exacerbations (excluding current exacerbation) within the previous year (exacerbation defined as: an event in the natural course of the disease characterized by a change in the patient's baseline dyspnea, cough and /or sputum beyond day to day variability sufficient to warrant a change in management of COPD (eg, treated with antibiotics and/or systemic corticosteroids or requiring an emergency room visit or an overnight stay at a hospital), OR
   2. Subject has had oxygen therapy use within 3 months prior to study entry.
2. Subject is a current or ex-smoker with at least 10 pack year smoking history (eg, at least 1 pack/day for 10 years, or equivalent).
3. Subject is willing and able to attend study visits/telephone contacts and adhere to all study assessments/procedures.
4. Subject is willing and able to provide written informed consent.

Exclusion Criteria:

1. Subject has current evidence or recent history of any clinically significant and unstable disease (other than COPD) or abnormality in the opinion of the Investigator that would put the subject at risk or which would compromise the quality of the study data; including but not limited to cardiovascular disease, myocardial infarction, cardiac failure, uncontrolled hypertension, life threatening arrhythmias, uncontrolled diabetes, neurologic or neuromuscular disease, liver disease, gastrointestinal disease or electrolyte abnormalities.
2. Subject has a primary diagnosis of asthma.
3. Subject has a history of tuberculosis, bronchiectasis or other non-specific pulmonary disease.
4. Subject has a history of urinary retention or bladder neck obstruction type symptoms.
5. Subject has a history of narrow angle glaucoma.
6. Subject has a recent history (previous 12 months) of excessive use or abuse of alcohol or narcotic/illegal drugs, as assessed by the Investigator.
7. Subject has a history of hypersensitivity or intolerance to aerosol medications, beta-2 agonists, or anticholinergics.
8. Subject is participating in another investigational drug study where drug was received within 30 days prior to Screening, or current participation in another investigational drug trial.
9. Subject is a staff member of the clinical site or a relative of a clinical site staff member.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-09-14 (Actual); Study Completion 2016-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Respiratory Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (28):
- United States (28):
  - Birmingham VA Medical Center, Birmingham, Alabama
  - Clinical Trial Connection, Flagstaff, Arizona
  - Waterbury Pulmonary Associates LLC, Waterbury, Connecticut
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Southeastern Intergrted Medical, PL d/b/a Florida Medical Research, Gainesville, Florida
  - Miami VA Medical Center, Miami, Florida
  - Gwinnett Biomedical Research, Lawrenceville, Georgia
  - University of Maryland Medical Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - VA Western New York Healthcare System, Buffalo, New York
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Gastonia Phannaceutical Research, Gastonia, North Carolina
  - Clinical Research of Lake Norman, Huntersville, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Cincinnati Veterans Affairs Medical Center, Cincinnati, Ohio
  - Remington-Davis, Inc., Columbus, Ohio
  - Consolidated Clinical Trials, Inc., Monroeville, Pennsylvania
  - Temple University Hospital, Temple Lung Center, Philadelphia, Pennsylvania
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - S. Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - Mid State Pulmonary, Nashville, Tennessee
  - Family Medicine Rural Health Clinic, PA, DBA FMC Science, Lampasas, Texas
  - Metroplex Pulmonary and Sleep Center, McKinney, Texas
  - Alamo Clinical Research Associates, San Antonio, Texas
  - Swedish Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Before recruitment and enrollment, each prospective subject was given a full explanation of the study, allowed to read the approved informed consent form and was provided ample time and the opportunity to ask any questions that may have arose.
Pre-assignment Details: Once all questions had been answered and the Investigator was assured that the prospective subject understood the implications of participating in the study, the prospective subject was asked to give consent to participate in the study by signing the informed consent form.
Period: Overall Study
Arm/Group | BROVANA | SPIRIVA
Started | 32 | 34
Completed | 23 | 31
Not Completed | 9 | 3
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — all other reasons combined | 2 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: full analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | BROVANA | SPIRIVA | Total
Number analyzed (Participants) | 32 | 34 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (6.86) | 72.1 (6.65) | 72.0 (6.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 14 | 18 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 32 | 34 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 26 | 27 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 34 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing All-cause Hospitalization or Emergency Department Visit Within 90-days of Initiating Treatment
Description: Due to early termination of the study, insufficient data were available to perform the statistical analyses described in the protocol. Only summary tables and listings, disposition, demographics, vital signs, AEs and listings of safety data were generated.
Time Frame: Up to 90 days
Population: Due to early termination of the study, insufficient data were available to perform the statistical analyses described in the protocol.
Arm/Group | BROVANA | SPIRIVA
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The AE reporting period lasts ~ 19 months
Arm/Group | BROVANA | SPIRIVA
All-Cause Mortality (participants affected / at risk) | 2/32 | 1/34
Serious Adverse Events (participants affected / at risk) | 15/32 | 13/34
Other Adverse Events (participants affected / at risk) | 19/32 | 23/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BROVANA (N=32) | SPIRIVA (N=34)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
cardia failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
death (General disorders) | 0 (0) | 1 (1)
acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 6 (6) | 0 (0)
pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
sepsis (Infections and infestations) | 0 (0) | 1 (1)
septic shock (Infections and infestations) | 1 (1) | 0 (0)
streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
blood testosterone decreased (Investigations) | 1 (1) | 0 (0)
hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 10 (13)
chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BROVANA (N=32) | SPIRIVA (N=34)
anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
artial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
dry eye (Eye disorders) | 0 (0) | 1 (1)
abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
consitpation (Gastrointestinal disorders) | 1 (1) | 4 (4)
diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
asthenia (General disorders) | 0 (0) | 2 (2)
chest discomfort (General disorders) | 2 (2) | 0 (0)
fatigue (General disorders) | 0 (0) | 3 (3)
generalised oedema (General disorders) | 0 (0) | 1 (1)
non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
odema peripheral (General disorders) | 0 (0) | 1 (1)
pyrexia (General disorders) | 1 (1) | 2 (3)
cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (2)
acute sinusitis (Infections and infestations) | 0 (0) | 2 (3)
bronchitis (Infections and infestations) | 0 (0) | 2 (2)
cellulitis (Infections and infestations) | 1 (1) | 1 (1)
oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
pneumonia (Infections and infestations) | 1 (1) | 0 (0)
sepsis (Infections and infestations) | 1 (1) | 0 (0)
sinusitis (Infections and infestations) | 1 (1) | 1 (1)
urinary tract infection (Infections and infestations) | 2 (2) | 1 (2)
arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (4)
wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1)
oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
troponin increased (Investigations) | 0 (0) | 1 (1)
white blood cell count increased (Investigations) | 0 (0) | 1 (1)
gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (5)
hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 2 (2) | 3 (3)
mental iimpairment (Nervous system disorders) | 1 (1) | 0 (0)
migraine (Nervous system disorders) | 1 (1) | 0 (0)
parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
confusional state (Psychiatric disorders) | 0 (0) | 2 (2)
delirium (Psychiatric disorders) | 0 (0) | 1 (1)
insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
renial failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 8 (9)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
study was terminated early due to lack of enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming with twenty-four (24) months following completion of the study at all sites, institution and investigator shall be free to publish.